CLINICAL TRIAL: NCT03709589
Title: Comparison of 7th Day All-Cause Mortality Among HDU Patients With Modified Early Warning Score of ≥ 5 With Those With Score of < 5
Brief Title: Comparison of Mortality Among HDU Patients With Modified Early Warning Score Cutoff of 5
Status: Completed | Type: Observational
Sponsor: Bader Faiyaz Zuberi (Other)
Responsible Party: Sponsor-Investigator, Bader Faiyaz Zuberi, Professor, Dow University of Health Sciences
Organization: Dow University of Health Sciences (Other)
Other Study IDs: MEWS-5
Record Dates: First submitted 2018-10-15; First posted 2018-10-17 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Critical Illness; Morality
Keywords: Mortality; High Dependency Unit; Modified Early Warning Score
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group-A: Patients with Modified Early Warning Score of ≥ 5
  Interventions: Other: Modified Early Warning Score
- Group-B: Patients with Modified Early Warning Score of < 5
  Interventions: Other: Modified Early Warning Score

INTERVENTIONS:
Other: Modified Early Warning Score — Modified Early Warning Score

SUMMARY:
Early categorization of critically ill patients by calculating MEWS score in hospitals may give a time window for appropriate steps. If a patient is suffering from sepsis, timely intravenous fluids, early antibiotics and monitoring in a low resource country like Pakistan, may have a great impact. Therefore, the current research is planned to early identify critically ill patients by applying MEWS and reducing the mortality by providing early management and taking appropriate life saving measures.

Objective: To compare frequency of mortality on 7th day of admission in HDU patients with Modified Early Warning Score at the time of admission of < 5 & ≥ 5.

DETAILED DESCRIPTION:
Early recognition and immediate resuscitation are fundamentals of successful management of all critically ill patients if they are suffering from infection and sepsis, malnutrition, AIDS, trauma, diabetes mellitus, drug overdose, and poisoning. In most, seriously ill patients, initial diagnosis may not be clear and immediate objective is to save the life and reverse or prevent vital organ damage e.g. brain, lungs, liver and kidneys. A rapid identifying, low cost method called as Modified Early Warning Score (MEWS) that utilize easy to measure physiological parameters such as vital signs and level of consciousness can be used to identify critical illness, facilitate early intervention and predict mortality. MEWS values range from 0 to maximum 14, higher scores mean greater hemodynamic instability. A score of 5 or more identifies a patient to be critically ill and is associated with increased risk of ICU admission and death. The negative predictive value of early warning MEWS < 3 was 98.1%, indicating the reliability of this score as a screening tool MEWS (modified early warning score) is a reliable screening tool to identify critically ill patients early and to act timely to improve outcomes in health care and prevent adverse events like cardiac arrest, renal failure. A study performed in Uganda on sepsis patients demonstrated that early IV fluid and antibiotic therapy together with vital sign monitoring was associated with lowered 30-day mortality.

Rationale: Early categorization of critically ill patients by calculating MEWS score in hospitals may give a time window for appropriate steps. If a patient is suffering from sepsis, timely intravenous fluids, early antibiotics and monitoring in a low resource country like Pakistan, may have a great impact. Therefore, the current research is planned to early identify critically ill patients by applying MEWS and reducing the mortality by providing early management and taking appropriate life saving measures.

ELIGIBILITY:
Inclusion Criteria:

* admitted in high dependency unit (HDU) of Medical Unit-II

Exclusion Criteria:

* Neurosurgical trauma clinically assessed
* Orthopedics or general surgery trauma patients clinically assessed
* Obstetrics patients clinically assessed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to HDU for any reason
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Mortality | 7 Days
  Status of Alive, Dead or Discharged on 7th Day

CONTACTS AND LOCATIONS:
Overall Officials: Bader F Zuberi, FPCS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Ruth KM Pauf Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathukia C, Fan W, Vadyak K, Biege C, Krishnamurthy M. Modified Early Warning System improves patient safety and clinical outcomes in an academic community hospital. J Community Hosp Intern Med Perspect. 2015 Apr 1;5(2):26716. doi: 10.3402/jchimp.v5.26716. eCollection 2015. PMID 25846353
- [Result] Nishijima I, Oyadomari S, Maedomari S, Toma R, Igei C, Kobata S, Koyama J, Tomori R, Kawamitsu N, Yamamoto Y, Tsuchida M, Tokeshi Y, Ikemura R, Miyagi K, Okiyama K, Iha K. Use of a modified early warning score system to reduce the rate of in-hospital cardiac arrest. J Intensive Care. 2016 Feb 9;4:12. doi: 10.1186/s40560-016-0134-7. eCollection 2016. PMID 26865981
- [Result] van Galen LS, Dijkstra CC, Ludikhuize J, Kramer MH, Nanayakkara PW. A Protocolised Once a Day Modified Early Warning Score (MEWS) Measurement Is an Appropriate Screening Tool for Major Adverse Events in a General Hospital Population. PLoS One. 2016 Aug 5;11(8):e0160811. doi: 10.1371/journal.pone.0160811. eCollection 2016. PMID 27494719
- [Result] Kruisselbrink R, Kwizera A, Crowther M, Fox-Robichaud A, O'Shea T, Nakibuuka J, Ssinabulya I, Nalyazi J, Bonner A, Devji T, Wong J, Cook D. Modified Early Warning Score (MEWS) Identifies Critical Illness among Ward Patients in a Resource Restricted Setting in Kampala, Uganda: A Prospective Observational Study. PLoS One. 2016 Mar 17;11(3):e0151408. doi: 10.1371/journal.pone.0151408. eCollection 2016. PMID 26986466